CLINICAL TRIAL: NCT05316259
Title: A Phase 1, Single-center, Open-Label, Randomized, 2 Period Crossover Study to Estimate the Effect of Food on the Pharmacokinetics of BPI-16350 in Chinese Healthy Volunteers After a Single Oral Administration
Brief Title: A Food-Effect Study of BPI-16350 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BTP-66732FE
Record Dates: First submitted 2022-03-14; First posted 2022-04-07 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A（Dosing in the fasted state followed by fed dosing） (Experimental): Dosing in the fasted state followed by fed dosing.A washout period of 14 days will be maintained between the 2 treatment periods.
  Interventions: Drug: BPI-16350
- Group B（Dosing in the fed state followed by fasted dosing） (Experimental): Dosing in the fed state followed by fasted dosing.A washout period of 14 days will be maintained between the 2 treatment periods.
  Interventions: Drug: BPI-16350

INTERVENTIONS:
Drug: BPI-16350 — Administered orally

SUMMARY:
This study is intended to quantify the effect of food on the pharmacokinetics of BPI-16350.

Subjects will be randomized to a crossover sequence at a 1:1 ratio and administered the dose of BPI-16350 on Day 1 in Period 1 and on Day 15 in Period 2 under fasting conditions(Treatment A) or with a high-fat meal(Treatment B).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 18~45 (including 18 and 45 years old);
* Male body weight ≥ 50kg, female body weight ≥ 45kg, body mass index (BMI) within the range of 19 ~ 26kg /m2;
* Clinical laboratory evaluations within the reference range for the test laboratory, unless deemed not clinically significant by the Investigator;
* The subjects should took effective contraceptive measures voluntarily from informed consent until 3 months after Study Completion；
* Able to comprehend and willing to sign an informed consent form.

Exclusion Criteria:

* History of significant hypersensitivity to any drug compound or food；
* Significant history or clinical manifestation of any significant cardiovascular, hepatic, renal, pulmonary, gastrointestinal, neurological, metabolic, musculoskeletal,hematological disorder；
* Hepatitis B virus surface antigen, hepatitis C virus antibody, treponema pallidum antibody or human immunodeficiency virus antibody is positive；
* Family history of long QTc syndrome; History or presence of an abnormal ECG；
* Drug abusers, smokers or alcoholics；
* Use of any medications within 14 days prior to the first administration；
* Donation of blood ≥ 200 mL or receipt of blood products within 3 months before enrollment, or plan on blood donation during the study period；
* Participation in any other investigational drug study or receive any vaccine within 3 months before enrollment；
* Female subjects who are pregnant or lactating；the serum HCG test of women with fertility is postive at Screening.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Cmax | from Day 1 to Day 9 after the first dose and from Day 15 to Day 23 after the second dose
  Maximum observed concentration
AUC0-t | from Day 1 to Day 9 after the first dose and from Day 15 to Day 23 after the second dose
  Area under the concentration-time curve from time 0 to time t
AUC0-∞ | from Day 1 to Day 9 after the first dose and from Day 15 to Day 23 after the second dose
  Area under the concentration-time curve from time 0 to infinity

SECONDARY OUTCOMES:
Tmax | from Day 1 to Day 9 after the first dose and from Day 15 to Day 23 after the second dose
  Time to reach maximum observed plasma concentration
t1/2 | from Day 1 to Day 9 after the first dose and from Day 15 to Day 23 after the second dose
  Half-life time
λz | from Day 1 to Day 9 after the first dose and from Day 15 to Day 23 after the second dose
  Elimination rate constant
tlag | from Day 1 to Day 9 after the first dose and from Day 15 to Day 23 after the second dose
  Lag Time
AUC %Extrap | from Day 1 to Day 9 after the first dose and from Day 15 to Day 23 after the second dose
  Percentage of AUCinf due to extrapolation from Tlast to infinity
CL/F | from Day 1 to Day 9 after the first dose and from Day 15 to Day 23 after the second dose
  Apparent Oral Clearance
V/F | from Day 1 to Day 9 after the first dose and from Day 15 to Day 23 after the second dose
  Apparent Volume of Distribution
Characterize the safety of BPI-16350 | from Day 1 to Day 23
  Number of subjects with treatment related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Haibin Yu, Ph.D, Principal Investigator — Kthics Committee (seal),of Beijing Youan Hospital,Capital Medical University
Locations (1):
- Kthics Committee (seal),of Beijing Youan Hospital,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No